CLINICAL TRIAL: NCT00169988
Title: Sertraline Alone vs. in Combination With Risperidone in the Treatment of Attenuated Positive and Negative Symptoms
Brief Title: Antidepressant and Antipsychotic to Treat Attenuated Positive and Negative Symptoms
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwell Health (Other)
Collaborators: Stanley Medical Research Institute (Other); Janssen Pharmaceutica N.V., Belgium (Industry); Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Diagnostic
Other Study IDs: 05-04-103
Record Dates: First submitted 2005-09-09; First posted 2005-09-15 (Estimated); Last update posted 2009-12-17 (Estimated); Status verified 2007-10

CONDITIONS: Prodromal Schizophrenia; Psychotic Disorders
Keywords: clinical high risk; attenuated positive symptoms; attenuated negative symptoms; cognition; functional status; prodromal psychosis
MeSH Terms: conditions — Schizotypal Personality Disorder; Psychotic Disorders | interventions — Risperidone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: risperidone
Drug: sertraline-primary

SUMMARY:
The Recognition and Prevention (RAP) Program is conducting a research study comparing an antidepressant, sertraline, alone versus in combination with a second-generation antipsychotic, risperidone, to evaluate their ability to reduce unusual thoughts, suspiciousness and other unusual experiences, to improve reasoning ability, memory, attention and social skills in adolescents.

DETAILED DESCRIPTION:
Eligible patients are enrolled in a 16-week trial consisting of symptom and side effects ratings (10 visits), monthly blood and urine tests, and neuropsychological testing at the first and last visits. At the initial appointment, all patients are assigned to sertraline and are randomly assigned to an adjunctive risperidone or placebo group. The treating physician is also blind to the medication assignment, which allows both the doctor and the patient to assess side effects and symptom improvement, unbiased by expectation. All patients receive an active medication.

ELIGIBILITY:
Inclusion Criteria:

* Participants are between the ages of 12 and 22.
* Participants are English-speaking.
* Participants are experiencing one or more symptoms like unusual thoughts, suspiciousness, or unusual perceptual experiences.
* Participants meet additional RAP criteria (evaluated during screening and interview).

Exclusion Criteria:

* Participants have been diagnosed with an Axis I psychotic disorder, including: schizophreniform disorder, schizophrenia, schizoaffective disorder, bipolar disorder, or major depression with psychotic features.
* Participants have a history of neurological, neuroendocrine, or other medical conditions known to affect the brain.
* Participants have a medical condition that contraindicates treatment with sertraline or risperidone.
* Participants have past or current substance dependence.
* Participants are currently taking and responding well to antidepressant or antipsychotic medication

Ages: 12 Years to 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 8 (Actual)
Dates: Start 2004-03; Study Completion 2007-04 (Actual)

PRIMARY OUTCOMES:
Score on attenuated positive symptom scale at 16 weeks
Score on attenuated negative symptom scale at 16 weeks

SECONDARY OUTCOMES:
Score on social functioning measure at 16 weeks
Score on academic functioning measure at 16 weeks
Score on cognitive measures at 16 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Barbara A Cornblatt, PhD, Principal Investigator — Long Island Jewish Medical Center (LIJMC); Christoph U Correll, MD, Study Director — LIJMC
Locations (1):
- RAP Program, Dept. of Psychiatry Research, The Zucker Hillside Hospital, Glen Oaks, New York, United States